CLINICAL TRIAL: NCT06641453
Title: Phase I/II Study of CAR-T Cell Therapy Targeting GPC3 in Patients with Treated Advanced GPC3-Positive Hepatocellular Carcinoma
Brief Title: CAR-T Cell Therapy Targeting GPC3 in Patients with Advanced GPC3-Positive Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of the Department of Biotherapeutics, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2024-560-01
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: HCC; GPC3; CAR-T cells
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GPC3 CAR-T cell therapy (Experimental): Enrolled patients will receive a single infusion of GPC3 CAR-T cells at a starting dose of 1×10^6 cells/kg.
  Interventions: Biological: GPC3-CART cells; Drug: Fludarabine Phosphate for Injection; Drug: Cyclophosphamide for Injection

INTERVENTIONS:
Biological: GPC3-CART cells — Phase 1: Dose escalation (3+3): Dose 1 (1 × 10^6 cells/kg) with or without FC regimen, Dose 2 (3 × 10^6 cells/kg), Dose 3 (6 × 10^6 cells/kg).
  Phase 2: Dose at RP2D.
Drug: Fludarabine Phosphate for Injection — Administered intravenously at a dose of 20-30 mg/m²/day on days -5, -4, and -3.
Drug: Cyclophosphamide for Injection — Administered intravenously at a dose of 300-500 mg/m²/day on days -5, -4, and -3.

SUMMARY:
In this single-center, single-arm, prospective, open-label Phase 1/2 study, the safety and efficacy of autologous GPC3-targeted chimeric antigen receptor (CAR) T-cell therapy will be evaluated in patients with GPC3-positive advanced hepatocellular carcinoma.

Phase 1 will involve the enrollment of six eligible patients to receive hepatic arterial infusion of GPC3-CAR T cells at a fixed dose of 1×10^6 cells/kg, with or without a standard lymphodepleting conditioning regimen (fludarabine and cyclophosphamide). Based on the results, it will be assessed whether the FC lymphodepletion regimen is necessary. Subsequently an additional six patients will be enrolled in a "3+3" dose-escalation design to adjust the dose of GPC3-CAR T cells to achieve optimal safety and efficacy. The recommended Phase 2 dose (RP2D) will then be established.

Phase 2 will involve the enrollment of 10-20 additional eligible patients to receive GPC3-CAR T cell therapy at the RP2D.

DETAILED DESCRIPTION:
Glypican-3 (GPC3) is a member of the glypican family, a group of heparan sulfate proteoglycans that are anchored to the cell membrane via a glycosylphosphatidylinositol (GPI) linkage. Structurally, GPC3 is composed of a core protein and covalently attached heparan sulfate chains. The core protein consists of an N-terminal domain, a large cysteine-rich region, and a C-terminal region that interacts with the cell membrane. Functionally, GPC3 is involved in regulating cell growth, differentiation, and apoptosis through interactions with various growth factors, including Wnt, Hedgehog, and fibroblast growth factors (FGFs). GPC3 plays a critical role during embryonic development but is largely absent in most adult tissues. However, its re-expression in certain cancers, particularly hepatocellular carcinoma (HCC), makes it an attractive target for therapeutic intervention.

GPC3 is highly and specifically expressed in hepatocellular carcinoma, a common form of primary liver cancer, while being minimally expressed in normal adult liver tissues. This differential expression makes GPC3 an appealing and specific target for cancer therapy.In HCC, GPC3 has been shown to play a role in promoting tumor growth and angiogenesis, enhancing tumor invasiveness, and protecting cancer cells from apoptosis. Due to its overexpression in HCC tumor tissues, GPC3 has been widely recognized as a potential biomarker for diagnosis, prognosis, and targeted therapies. Its selective expression in cancerous tissue with limited distribution in normal tissues makes it an ideal candidate for chimeric antigen receptor (CAR) T cell therapy, which aims to specifically target and destroy cancer cells while minimizing off-target effects.

Several studies have explored the use of GPC3-targeted CAR T cell therapies in hepatocellular carcinoma. These early clinical trials were designed to evaluate the safety and preliminary efficacy of GPC3-CAR T cell treatments in patients with advanced-stage, GPC3-positive HCC. The results from these trials demonstrated that GPC3-CAR T cell therapy is generally safe, with manageable adverse effects, and some patients exhibited clinical responses, such as tumor regression or disease stabilization. However, despite these promising results, the overall efficacy of GPC3-CAR T cell therapy did not meet the threshold required for routine clinical application. The responses were often transient, and relapse occurred in many patients due to challenges such as T cell exhaustion, limited CAR T cell persistence, and the immunosuppressive tumor microenvironment (TME) associated with HCC. These limitations highlighted the need for further optimization of the CAR T cell design and administration strategies to improve the efficiency of GPC3-targeted therapies in HCC.

Building on the foundation of these earlier studies, the investigators aim to conduct a prospective, open-label, phase 1/2 clinical trial to evaluate our newly optimized GPC3-targeted CAR T cell therapy in patients with advanced-stage, GPC3-positive HCC. Our approach introduces two major innovations compared to previous studies:

1. Novel CAR T Cell Design Strategy: In addition to the traditional CAR structure comprising a single-chain variable fragment (scFv) specific for GPC3, a co-stimulatory domain (41BB/CD28), and a CD3ζ activation domain, we have incorporated novel immune microenvironment-activating elements. These elements are designed to enhance the activation and proliferation of CAR T cells while simultaneously recruiting and activating antigen-presenting cells (APCs) and bystander immune effector cells. This dual activation strategy aims to overcome the immunosuppressive TME and promote a more robust and sustained anti-tumor response.
2. New Administration Route: Unlike previous studies that primarily used intravenous administration, the investigators have developed a new method of delivering CAR T cells directly into the tumor site. This strategy is intended to facilitate immediate and direct contact between the CAR T cells and the tumor cells, allowing for more efficient tumor infiltration and modification of the TME. By altering the local immune landscape, the investigators aim to enhance CAR T cell persistence and efficacy while reducing the likelihood of tumor escape.

By leveraging these two innovative strategies, the investigators aim to achieve improved clinical outcomes in terms of both safety and efficacy. The investigators hypothesize that the inclusion of immune microenvironment-activating elements will enhance the activation of not only CAR T cells but also the broader immune system, creating a more hostile environment for tumor cells. Furthermore, direct tumor delivery of CAR T cells may increase their local concentration and activity, reducing the tumor burden more effectively. Through this optimized approach, the investigators hope to provide a more potent and durable therapeutic option for patients with GPC3-positive hepatocellular carcinoma, addressing the limitations encountered in previous trials.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70 years old (inclusive); gender unrestricted.

Diagnosis of advanced Hepatocellular Carcinoma (HCC), meeting the following requirements:

* Pathologically Confirmed: Diagnosis of HCC confirmed by histopathology. Staging: Classified as China Liver Cancer (CNLC) stage IIb-IIIb, having undergone treatments recommended by the "Primary Liver Cancer Diagnosis and Treatment Guidelines (2024 Edition)" with disease progression and either no further recommended treatments available or intolerance to the recommended treatment options.
* Measurable Lesion: At least one measurable lesion as defined by RECIST v1.1 criteria.
* Tumor Sample Availability: Availability of tumor tissue samples or samples obtained by tumor biopsy for GPC3 expression quantification and other related analyses.
* GPC3 Positivity: Confirmed positive GPC3 expression by immunohistochemistry (IHC), where positivity is defined as a quantified immunohistochemical score of "+" or above.
* ECOG Performance Status: Eastern Cooperative Oncology Group (ECOG) score of 0-1.
* Life Expectancy: Expected survival time of ≥ 3 months.
* Cirrhosis Status: Child-Pugh class A or B for liver cirrhosis.
* Organ Function: Must meet the following organ function requirements:

Hematology:

Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L (no granulocyte colony-stimulating factor support within 7 days prior to testing).

Absolute lymphocyte count (ALC) ≥ 0.5 × 10^9/L; hemoglobin (HGB) ≥ 80 g/L (no red blood cell transfusion within 7 days prior to testing).

Platelet count (PLT) ≥ 75 × 10^9/L (no transfusion support within 7 days prior to testing).

Liver Function:

Aspartate aminotransferase (AST ) and alanine aminotransferase (ALT ) ≤ 3.0 × upper limit of normal (ULN).

Total bilirubin (TBIL) ≤ 2.0 × ULN (≤ 3.0 × ULN for patients with Gilbert's syndrome and direct bilirubin ≤ 1.5 × ULN).

Coagulation Function:

International normalized ratio (INR) ≤ 1.5 × ULN. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (except for patients receiving therapeutic anticoagulants).

Renal Function: Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min.

Cardiac Function: Left ventricular ejection fraction (LVEF) ≥ 50% (confirmed by echocardiography).

Pulmonary Function: Pulse oxygen saturation (SpO2) > 93% at rest without supplemental oxygen.

* Contraception: Women of childbearing potential must have a negative pregnancy test, and both male and female participants with reproductive potential must agree to use effective contraception throughout the screening and study period until one year after the last cellular infusion.
* Informed Consent: Willingness to provide voluntary written informed consent and compliance with the study protocol.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Positive HCV RNA quantification, positive human immunodeficiency virus (HIV) antibodies, or active syphilis infection.
* Chronic HBV infection with serum HBV-DNA levels ≥ 500 IU/mL.
* Unresolved non-hematologic toxicities (excluding alopecia and peripheral sensory neuropathy) from prior treatments (surgery, chemotherapy, radiotherapy, targeted therapy, immunotherapy) that have not improved to ≤ Grade 1 according to CTCAE.
* History of allogeneic tissue/organ transplantation (including bone marrow, stem cell, liver, or kidney transplants), except those that do not require immunosuppressive therapy (e.g., corneal or hair transplants).
* Prior treatment targeting GPC3.
* Receipt of anti-tumor treatment for liver cancer or any other medical intervention that could impair major organ function within four weeks before signing informed consent.
* Known central nervous system metastasis.
* Presence of clinically significant systemic disease (e.g., severe active - - infections, significant heart, lung, liver, kidney, or neurological dysfunction) that, in the investigator's opinion, may impair the patient's ability to tolerate the study treatment or increase the risk of complications. Including but not limited to:

  1. Uncontrolled severe active infection.
  2. Symptomatic congestive heart failure (NYHA Class II-IV).
  3. Clinically significant severe aortic valve stenosis or symptomatic mitral valve stenosis.
  4. QTc > 450 msec on ECG, or QTc > 480 msec in patients with bundle branch block.
  5. Uncontrolled clinically significant arrhythmias within six months before signing informed consent.
  6. Acute coronary syndrome (e.g., unstable angina or myocardial infarction) within six months before signing informed consent.
  7. Hypertension not controlled by medication (systolic BP ≥ 160 mmHg and/or diastolic BP ≥ 100 mmHg).
  8. Cerebrovascular accidents, including transient ischemic attack (TIA), cerebral infarction, cerebral hemorrhage, or subarachnoid hemorrhage within six months before signing informed consent.
  9. Active, chronic, or recurrent severe autoimmune disease (within one year before signing informed consent), or liver cirrhosis/liver cancer caused by autoimmune hepatitis.
  10. Any form of primary or secondary immunodeficiency, such as severe combined immunodeficiency (SCID).
  11. Risk of organ perforation or hemorrhage, as determined by the investigator.
* History of severe systemic hypersensitivity to study drugs/components [e.g., fludarabine, cyclophosphamide, dimethyl sulfoxide (DMSO), low molecular weight dextran, human serum albumin (HSA)].
* Receipt of live attenuated vaccine within four weeks before signing informed consent.
* Participation in another clinical trial within four weeks before signing informed consent.
* History of another malignancy within the past five years, excluding adequately treated non-melanoma skin cancer or carcinoma in situ (e.g., breast, stomach, colon, bladder, cervix, or melanoma).
* History of neuropsychiatric disorders diagnosed by ICD-11 criteria, or any neuropsychiatric disorder deemed by the investigator to warrant exclusion, including but not limited to epilepsy, schizophrenia, dementia, or addiction to drugs/alcohol.
* Any other condition that, in the investigator's opinion, makes the patient unsuitable for this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | Up to 12 months since the initiation of GPC3-targeted CAR T cell therapy.
  Treatment-related adverse events are defined as any medical events occurring since the initiation of GPC3-targeted CAR T cell therapy. CRS or CRES will be graded based on the American Society for Transplantation and Cellular Therapy (ASTCT) criteria, and other adverse events will be graded according to CTCAE v5.0.
Incidence of dose-limiting toxicities (DLTs) | Up to 28 days from the initiation of GPC3-targeted CAR T cell therapy.
  Dose-limiting toxicities are defined as GPC3-targeted CAR T cell therapy-related adverse events within the first 28 days that meet the following criteria: grade 3 or higher CRS or CRES, and any other grade 4 adverse events.

SECONDARY OUTCOMES:
Number and copy number of GPC3-targeted CAR T cells | Up to 3 years from the initiation of GPC3-targeted CAR T cell therapy.
  The number and copy number of GPC3-targeted CAR T cells are evaluated in peripheral blood and tumor tissue.
Objective response rate (ORR) | Up to 3 years from the initiation of GPC3-targeted CAR T cell therapy.
  Objective response rate includes complete response and partial response, as defined by investigators according to RECIST 1.1 criteria.
Progression Free Survival (PFS) | Up to 3 years from the initiation of GPC3-targeted CAR T cell therapy.
  Progression Free Survival is defined as the time from the initiation of GPC3 targeted CAR T cell therapy to documented disease progression or death.
Time to response (TTR) | Up to 3 years from the initiation of GPC3-targeted CAR T cell therapy.
  TTR is defined as the time from the initiation of GPC3 targeted CAR T cell therapy to first assessed CR or PR by investigators according to RECIST 1.1 criteria.
Duration of response (DOR) | Up to 3 years from the initiation of GPC3-targeted CAR T cell therapy.
  Duration of response is defined as the time from objective response until documented tumor progression among responders.
Overall Survival (OS) | Up to 3 years from the initiation of GPC3-targeted CAR T cell therapy.
  Overall Survival is defined as the time from the initiation of GPC3 targeted CAR T cell therapy to documented disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Yangbin Zhao, Ph.D., Study Director — UTC Therapeutics Inc.
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided